CLINICAL TRIAL: NCT00030290
Title: Feasibility Study for Organ Confined Prostate Cancer Treatment With HIFU Using SONABLATE System
Brief Title: Ultrasound in Treating Patients With Prostate Cancer Confined to the Prostate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Focus Surgery (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: FOCUS-G000276; CDR0000069126 (Registry Identifier: PDQ (Physician Data Query)); CWRU-050130; IUMC-010233; NCI-V01-1684
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-12

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation

INTERVENTIONS:
Procedure: high-intensity focused ultrasound ablation

SUMMARY:
RATIONALE: Highly focused ultrasound energy may be able to kill cancer cells by heating the tumor without affecting the surrounding tissue.

PURPOSE: Phase I trial to study the effectiveness of focused ultrasound energy in treating patients who have prostate cancer that has not spread beyond the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of Sonablate to focus ultrasonic waves for the purpose of selectively destroying prostate cancer tissue, with resultant drop in PSA levels to below 0.5 ng/mL and negative biopsy for cancer cells, in patients with organ-confined prostate cancer.

OUTLINE: This is a multicenter study.

A probe is inserted into the rectum. High-intensity focused ultrasound (HIFU) energy using the Sonablate system is delivered to the prostate tissue over approximately 2-3 hours. Patients with residual cancer lesion (by biopsy), PSA greater than 0.5 ng/mL or increasing PSA levels taken at least 2 months apart, visible prostate tissue on ultrasound, and no local or distant metastases after day 90 undergo retreatment with HIFU.

Patients are followed at 2, 14, 30, 90, and 180 days.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed organ-confined prostate cancer (clinical stage T1 or T2 only)
* Pretreatment prostate weight less than 40 g
* Gleason score no greater than 7
* PSA no greater than 10 ng/mL
* No significant intravesical median lobe (greater than 2 cm) on ultrasound
* Able to visualize prostate gland adequately on transrectal ultrasound imaging
* No prostate calcification greater than 5 mm
* No metastases by bone scan

PATIENT CHARACTERISTICS:

Age:

* 40 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No bleeding disorder as determined by abnormal PT and PTT

Renal:

* No active urinary tract infection
* No history of urinary bladder neck contracture

Other:

* No prior allergy to latex
* No Anesthesia Surgical Assignment category IV or greater
* No interest in future fertility
* No history of inflammatory bowel disease
* No other concurrent major debilitating illness
* No other prior or concurrent malignancy except skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for prostate cancer

Chemotherapy:

* No prior chemotherapy for prostate cancer

Endocrine therapy:

* At least 3 months since prior hormonal therapy (including finasteride) for prostate cancer

Radiotherapy:

* No prior radiotherapy for prostate cancer

Surgery:

* No prior transurethral resection of prostate
* No prior urethral stent
* No prior major rectal surgery

Other:

* No prior cryotherapy for prostate cancer
* No prior thermotherapy
* No other prior therapy for prostate cancer
* No concurrent warfarin or other anticoagulant

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael O. Koch, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States